CLINICAL TRIAL: NCT03006575
Title: A Prospective, Randomized, Phase Ⅱ Study of Split-course Chemoradiotherapy For Locoregional Recurrence Of Non-small Cell Lung Cancer After Surgical Resection
Brief Title: Study of Split-course Chemoradiotherapy For Postoperative Locoregional Recurrence Of Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1017
Record Dates: First submitted 2016-04-13; First posted 2016-12-30 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Split-course Chemoradiotherapy; Locoregional recurrence; Postoperative recurrence
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

ARMS (1):
- split-course radiotherapy (Experimental): The radiotherapy is delivered using simultaneous integrated boost (SIB)-IMRT. Patients are irradiation at a palliative dose at the initial course: 40-51Gy/10-17f to PTV-GTV. The disease is re-evaluated one month after the end of the initial course using CT. The patient who achieved a partial remission according to the RECIST criteria and had a recovery of lung function should get the additional boost. At the second course, the tumor is repositioned and scanned. The residual tumor was then treated with the second course of radiotherapy. A dose of 15-24 Gy/5-8f is delivered to the residue tumor. Concurrent chemotherapy consists of weekly docetaxel(25mg/㎡) and nedaplatin(25mg/㎡), each of 1 day's duration.
  Interventions: Radiation: split-course radiotherapy; Drug: concurrent chemotherapy

INTERVENTIONS:
Radiation: split-course radiotherapy — split-course chest radiation at 40-51 Gy/10-17f and 15-24 Gy/5-8f
Drug: concurrent chemotherapy — weekly docetaxel(25mg/㎡) and nedaplatin(25mg/㎡) concurrent with chest radiation

SUMMARY:
This Phase II randomized study is to determine the efficacy of split-course irradiation with concurrent chemotherapy in locoregional recurrence of non-small cell lung cancer after surgical resection

DETAILED DESCRIPTION:
This Phase II randomized study is to determine the efficacy of split-course irradiation with concurrent chemotherapy in locoregional recurrence of non-small cell lung cancer after surgical resection.

Patients received four cycles of weekly docetaxel(25mg/㎡) and nedaplatin(25mg/㎡), each of 1 day's duration, combined with split-course thoracic radiotherapy of 40-51 Gy/10-17 fractions and 15-24 Gy/5-8 fractions administered in the first and second courses, respectively, with one-month break. The primary end point is progression-free survival, which is the time that passes from the first day of radiotherapy to the date at which disease progresses. Progression-free survival will be calculated using the Kaplan-Meier method.Toxicities will be graded according to CTCAE v. 4.0.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of NSCLC.
* Patients have measurable or evaluable lesions based on the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Postoperative locoregional recurrence including ipsilateral hemithorax and the mediastinum.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Previously treated with chemotherapy or treatment-naive
* No previous chest radiotherapy, immunotherapy or biotherapy
* Hemoglobin≥10 mg/dL, platelet≥100000/μL,absolute neutrophil count ≥1500/μL
* Serum creatinine ≤1.25 times the upper normal limit(UNL), or creatinine clearance≥60 ml/min
* Bilirubin ≤1.5 times UNL, AST（SGOT）≤2.5 times UNL ,ALT（SGPT）≤2.5 times UNL,alkaline phosphatase ≤5 times UNL
* Forced expiratory volume at one second (FEV1) >0.8 L
* Coagulation tests within normal limits
* patients and their family signed the informed consents

Exclusion Criteria:

* Previous or recent another malignancy, except nonmelanoma skin cancer or cervical cancer in situ
* Second primary carcinoma of the lung
* Contraindication for chemotherapy
* Malignant pleural or pericardial effusion.
* Women in pregnancy, lactation period, or no pregnancy test 14 days before the first dos
* Women who has the probability of pregnancy without contraception
* Tendency of hemorrhage
* In other clinical trials within 30 days
* Addicted in drugs or alcohol, AIDS patients
* Uncontrollable seizure or psychotic patients without self-control ability
* Severe allergy or idiosyncrasy
* Not suitable for this study judged by researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 2 years

SECONDARY OUTCOMES:
Overall Survival | 2 years
Response Rate | 2 years
rate of patients who develop local recurrence or distant recurrence | 2 year
rate of grade 3-4 radiation pneumonitis/esophagitis evaluated by Common Terminology Criteria for Adverse Events Version 4.0 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, professor, Principal Investigator — Sun yat-sen universtiy cancer center
Locations (1):
- Hui Liu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goldstraw P, Crowley J, Chansky K, Giroux DJ, Groome PA, Rami-Porta R, Postmus PE, Rusch V, Sobin L; International Association for the Study of Lung Cancer International Staging Committee; Participating Institutions. The IASLC Lung Cancer Staging Project: proposals for the revision of the TNM stage groupings in the forthcoming (seventh) edition of the TNM Classification of malignant tumours. J Thorac Oncol. 2007 Aug;2(8):706-14. doi: 10.1097/JTO.0b013e31812f3c1a. PMID 17762336
- [Background] Hung JJ, Hsu WH, Hsieh CC, Huang BS, Huang MH, Liu JS, Wu YC. Post-recurrence survival in completely resected stage I non-small cell lung cancer with local recurrence. Thorax. 2009 Mar;64(3):192-6. doi: 10.1136/thx.2007.094912. PMID 19252018
- [Background] Hung JJ, Jeng WJ, Hsu WH, Wu KJ, Chou TY, Hsieh CC, Huang MH, Liu JS, Wu YC. Prognostic factors of postrecurrence survival in completely resected stage I non-small cell lung cancer with distant metastasis. Thorax. 2010 Mar;65(3):241-5. doi: 10.1136/thx.2008.110825. PMID 20335294
- [Background] Williams BA, Sugimura H, Endo C, Nichols FC, Cassivi SD, Allen MS, Pairolero PC, Deschamps C, Yang P. Predicting postrecurrence survival among completely resected nonsmall-cell lung cancer patients. Ann Thorac Surg. 2006 Mar;81(3):1021-7. doi: 10.1016/j.athoracsur.2005.09.020. PMID 16488713
- [Background] Endo C, Sakurada A, Notsuda H, Noda M, Hoshikawa Y, Okada Y, Kondo T. Results of long-term follow-up of patients with completely resected non-small cell lung cancer. Ann Thorac Surg. 2012 Apr;93(4):1061-8. doi: 10.1016/j.athoracsur.2012.01.004. Epub 2012 Mar 3. PMID 22386090
- [Background] Hung JJ, Jeng WJ, Hsu WH, Chou TY, Huang BS, Wu YC. Predictors of death, local recurrence, and distant metastasis in completely resected pathological stage-I non-small-cell lung cancer. J Thorac Oncol. 2012 Jul;7(7):1115-23. doi: 10.1097/JTO.0b013e31824cbad8. PMID 22592210
- [Background] Sugimura H, Nichols FC, Yang P, Allen MS, Cassivi SD, Deschamps C, Williams BA, Pairolero PC. Survival after recurrent nonsmall-cell lung cancer after complete pulmonary resection. Ann Thorac Surg. 2007 Feb;83(2):409-17; discussioin 417-8. doi: 10.1016/j.athoracsur.2006.08.046. PMID 17257962
- [Background] Ichinose Y, Yano T, Yokoyama H, Inoue T, Asoh H, Tayama K, Takanashi N. Postrecurrent survival of patients with non-small-cell lung cancer undergoing a complete resection. J Thorac Cardiovasc Surg. 1994 Jul;108(1):158-61. PMID 8028360
- [Background] Saisho S, Yasuda K, Maeda A, Yukawa T, Okita R, Hirami Y, Shimizu K, Nakata M. Post-recurrence survival of patients with non-small-cell lung cancer after curative resection with or without induction/adjuvant chemotherapy. Interact Cardiovasc Thorac Surg. 2013 Feb;16(2):166-72. doi: 10.1093/icvts/ivs450. Epub 2012 Nov 9. PMID 23143203
- [Background] Yano T, Okamoto T, Fukuyama S, Maehara Y. Therapeutic strategy for postoperative recurrence in patients with non-small cell lung cancer. World J Clin Oncol. 2014 Dec 10;5(5):1048-54. doi: 10.5306/wjco.v5.i5.1048. PMID 25493240
- [Background] Green N, Kern W. The clinical course and treatment results of patients with postresection locally recurrent lung cancer. Cancer. 1978 Nov;42(5):2478-82. doi: 10.1002/1097-0142(197811)42:53.0.co;2-q. PMID 214222
- [Background] Yano T, Hara N, Ichinose Y, Asoh H, Yokoyama H, Ohta M, Hata K. Local recurrence after complete resection for non-small-cell carcinoma of the lung. Significance of local control by radiation treatment. J Thorac Cardiovasc Surg. 1994 Jan;107(1):8-12. PMID 8283923
- [Background] Kelsey CR, Marks LB, Hollis D, Hubbs JL, Ready NE, D'Amico TA, Boyd JA. Local recurrence after surgery for early stage lung cancer: an 11-year experience with 975 patients. Cancer. 2009 Nov 15;115(22):5218-27. doi: 10.1002/cncr.24625. PMID 19672942
- [Background] Feld R, Rubinstein LV, Weisenberger TH. Sites of recurrence in resected stage I non-small-cell lung cancer: a guide for future studies. J Clin Oncol. 1984 Dec;2(12):1352-8. doi: 10.1200/JCO.1984.2.12.1352. PMID 6512581
- [Background] Martini N, Bains MS, Burt ME, Zakowski MF, McCormack P, Rusch VW, Ginsberg RJ. Incidence of local recurrence and second primary tumors in resected stage I lung cancer. J Thorac Cardiovasc Surg. 1995 Jan;109(1):120-9. doi: 10.1016/S0022-5223(95)70427-2. PMID 7815787
- [Background] Kelsey CR, Clough RW, Marks LB. Local recurrence following initial resection of NSCLC: salvage is possible with radiation therapy. Cancer J. 2006 Jul-Aug;12(4):283-8. doi: 10.1097/00130404-200607000-00006. PMID 16925972
- [Background] Kasprzyk M, Slawinski G, Musik M, Marciniak L, Dyszkiewicz W, Piwkowski C, Galecki B. Completion pneumonectomy and chemoradiotherapy as treatment options in local recurrence of non-small-cell lung cancer. Kardiochir Torakochirurgia Pol. 2015 Mar;12(1):18-25. doi: 10.5114/kitp.2015.50563. Epub 2015 Mar 31. PMID 26336473
- [Background] Bar J, Ng D, Moretto P, Goss GD, Sun A, Macrae R, Laurie SA, Leighl N, Nicholas G. Chemoradiotherapy for locoregional recurrence of non-small-cell lung cancer after surgical resection: a retrospective analysis. Clin Lung Cancer. 2013 Mar;14(2):200-4. doi: 10.1016/j.cllc.2012.05.008. Epub 2012 Aug 4. PMID 22868221
- [Background] Curran WJ, Scott C, Langer C, et al. Phase III comoarision of sequential vs concurrent chemoradiation therapy for patients with unresectable stage III non-small cell lung cancer: initial report of RTOG 9410. Proc Am Soc Clin Oncol, 2000, 19: 484a.
- [Background] Furuse K, Fukuoka M, Kawahara M, Nishikawa H, Takada Y, Kudoh S, Katagami N, Ariyoshi Y. Phase III study of concurrent versus sequential thoracic radiotherapy in combination with mitomycin, vindesine, and cisplatin in unresectable stage III non-small-cell lung cancer. J Clin Oncol. 1999 Sep;17(9):2692-9. doi: 10.1200/JCO.1999.17.9.2692. PMID 10561343
- [Background] Auperin A, Le Pechoux C, Rolland E, Curran WJ, Furuse K, Fournel P, Belderbos J, Clamon G, Ulutin HC, Paulus R, Yamanaka T, Bozonnat MC, Uitterhoeve A, Wang X, Stewart L, Arriagada R, Burdett S, Pignon JP. Meta-analysis of concomitant versus sequential radiochemotherapy in locally advanced non-small-cell lung cancer. J Clin Oncol. 2010 May 1;28(13):2181-90. doi: 10.1200/JCO.2009.26.2543. Epub 2010 Mar 29. PMID 20351327
- [Background] Pfister DG, Johnson DH, Azzoli CG, Sause W, Smith TJ, Baker S Jr, Olak J, Stover D, Strawn JR, Turrisi AT, Somerfield MR; American Society of Clinical Oncology. American Society of Clinical Oncology treatment of unresectable non-small-cell lung cancer guideline: update 2003. J Clin Oncol. 2004 Jan 15;22(2):330-53. doi: 10.1200/JCO.2004.09.053. Epub 2003 Dec 22. No abstract available. PMID 14691125
- [Background] Shukuya T, Yamanaka T, Seto T, et al. Randomized phase III study of nedaplatin (N) plus docetaxel (D) versus cisplatin (C) plus D for advanced or relapsed squamous cell carcinoma of the lung (SqLC): WJOG5208L. Journal of Clinical Oncology, 2015 ASCO Annual Meeting (May 29 - June 2, 2015) Vol 33, No 15_suppl (May 20 Supplement), 2015: 8004
- [Background] Blackstock AW, Socinski MA, Bogart J, et al; Cancer and Leukemia Group B. Induction plus concurrent chemotherapy with high-dose (74 Gy) 3-dimensional (3-D) thoracic radiotherapy in stage III non-small cell lung cancer. Preliminary report of Cancer and Leukemia Group B (CALGB) 30105. Proc Am Soc Clin Oncol 2006;24(18S):Abstr 7042.
- [Background] Lee CB, Socinski A, Lin L, et al. High-dose 3D chemoradiotherapy in stage III non-small cell lung cancer (NSCLC) at the University of North Carolina: long-term follow up and late complications. Proc Am Soc Clin Oncol 2006;24(18S):Abstr 7145.
- [Background] Kong FM, Ten Haken RK, Schipper MJ, Sullivan MA, Chen M, Lopez C, Kalemkerian GP, Hayman JA. High-dose radiation improved local tumor control and overall survival in patients with inoperable/unresectable non-small-cell lung cancer: long-term results of a radiation dose escalation study. Int J Radiat Oncol Biol Phys. 2005 Oct 1;63(2):324-33. doi: 10.1016/j.ijrobp.2005.02.010. PMID 16168827
- [Background] Schild SE, McGinnis WL, Graham D, Hillman S, Fitch TR, Northfelt D, Garces YI, Shahidi H, Tschetter LK, Schaefer PL, Adjei A, Jett J. Results of a Phase I trial of concurrent chemotherapy and escalating doses of radiation for unresectable non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2006 Jul 15;65(4):1106-11. doi: 10.1016/j.ijrobp.2006.02.046. Epub 2006 May 26. PMID 16730134
- [Background] Bradley JD, Paulus R, Komaki R, Masters G, Blumenschein G, Schild S, Bogart J, Hu C, Forster K, Magliocco A, Kavadi V, Garces YI, Narayan S, Iyengar P, Robinson C, Wynn RB, Koprowski C, Meng J, Beitler J, Gaur R, Curran W Jr, Choy H. Standard-dose versus high-dose conformal radiotherapy with concurrent and consolidation carboplatin plus paclitaxel with or without cetuximab for patients with stage IIIA or IIIB non-small-cell lung cancer (RTOG 0617): a randomised, two-by-two factorial phase 3 study. Lancet Oncol. 2015 Feb;16(2):187-99. doi: 10.1016/S1470-2045(14)71207-0. Epub 2015 Jan 16. PMID 25601342
- [Background] Spoelstra FO, Pantarotto JR, van Sornsen de Koste JR, Slotman BJ, Senan S. Role of adaptive radiotherapy during concomitant chemoradiotherapy for lung cancer: analysis of data from a prospective clinical trial. Int J Radiat Oncol Biol Phys. 2009 Nov 15;75(4):1092-7. doi: 10.1016/j.ijrobp.2008.12.027. Epub 2009 Mar 26. PMID 19327915
- [Background] Gielda BT, Marsh JC, Zusag TW, Faber LP, Liptay M, Basu S, Warren WH, Fidler MJ, Batus M, Abrams RA, Bonomi P. Split-course chemoradiotherapy for locally advanced non-small cell lung cancer: a single-institution experience of 144 patients. J Thorac Oncol. 2011 Jun;6(6):1079-86. doi: 10.1097/JTO.0b013e3182199a7c. PMID 21532501
- [Background] Belani CP, Choy H, Bonomi P, Scott C, Travis P, Haluschak J, Curran WJ Jr. Combined chemoradiotherapy regimens of paclitaxel and carboplatin for locally advanced non-small-cell lung cancer: a randomized phase II locally advanced multi-modality protocol. J Clin Oncol. 2005 Sep 1;23(25):5883-91. doi: 10.1200/JCO.2005.55.405. Epub 2005 Aug 8. PMID 16087941
- [Background] Curran W, Scott C, Langer C, et al. Phase III comparison of sequential vs concurrent chemoradiotherapy for patients (pts) with unresected stage III non-small cell lung cancer (NSCLC): report of Radiation Therapy Oncology Group (RTOG) 9410. Proc Am Soc Clin Oncol 2003;22:Abstr 2499.
- [Background] Albain KS, Swann RS, Rusch VW, Turrisi AT 3rd, Shepherd FA, Smith C, Chen Y, Livingston RB, Feins RH, Gandara DR, Fry WA, Darling G, Johnson DH, Green MR, Miller RC, Ley J, Sause WT, Cox JD. Radiotherapy plus chemotherapy with or without surgical resection for stage III non-small-cell lung cancer: a phase III randomised controlled trial. Lancet. 2009 Aug 1;374(9687):379-86. doi: 10.1016/S0140-6736(09)60737-6. Epub 2009 Jul 24. PMID 19632716
- [Background] Vokes EE, Herndon JE 2nd, Kelley MJ, Cicchetti MG, Ramnath N, Neill H, Atkins JN, Watson DM, Akerley W, Green MR; Cancer and Leukemia Group B. Induction chemotherapy followed by chemoradiotherapy compared with chemoradiotherapy alone for regionally advanced unresectable stage III Non-small-cell lung cancer: Cancer and Leukemia Group B. J Clin Oncol. 2007 May 1;25(13):1698-704. doi: 10.1200/JCO.2006.07.3569. Epub 2007 Apr 2. PMID 17404369
- [Background] Hanna N, Neubauer M, Yiannoutsos C, McGarry R, Arseneau J, Ansari R, Reynolds C, Govindan R, Melnyk A, Fisher W, Richards D, Bruetman D, Anderson T, Chowhan N, Nattam S, Mantravadi P, Johnson C, Breen T, White A, Einhorn L; Hoosier Oncology Group; US Oncology. Phase III study of cisplatin, etoposide, and concurrent chest radiation with or without consolidation docetaxel in patients with inoperable stage III non-small-cell lung cancer: the Hoosier Oncology Group and U.S. Oncology. J Clin Oncol. 2008 Dec 10;26(35):5755-60. doi: 10.1200/JCO.2008.17.7840. Epub 2008 Nov 10. PMID 19001323
- [Background] Davies AM, Chansky K, Lau DH, Leigh BR, Gaspar LE, Weiss GR, Wozniak AJ, Crowley JJ, Gandara DR; SWOG S9712. Phase II study of consolidation paclitaxel after concurrent chemoradiation in poor-risk stage III non-small-cell lung cancer: SWOG S9712. J Clin Oncol. 2006 Nov 20;24(33):5242-6. doi: 10.1200/JCO.2006.07.0268. PMID 17114656
- [Background] Fu KK, Pajak TF, Trotti A, Jones CU, Spencer SA, Phillips TL, Garden AS, Ridge JA, Cooper JS, Ang KK. A Radiation Therapy Oncology Group (RTOG) phase III randomized study to compare hyperfractionation and two variants of accelerated fractionation to standard fractionation radiotherapy for head and neck squamous cell carcinomas: first report of RTOG 9003. Int J Radiat Oncol Biol Phys. 2000 Aug 1;48(1):7-16. doi: 10.1016/s0360-3016(00)00663-5. PMID 10924966
- [Background] Saunders M, Dische S, Barrett A, Harvey A, Griffiths G, Palmar M. Continuous, hyperfractionated, accelerated radiotherapy (CHART) versus conventional radiotherapy in non-small cell lung cancer: mature data from the randomised multicentre trial. CHART Steering committee. Radiother Oncol. 1999 Aug;52(2):137-48. doi: 10.1016/s0167-8140(99)00087-0. PMID 10577699
- [Background] Petereit DG, Sarkaria JN, Chappell R, Fowler JF, Hartmann TJ, Kinsella TJ, Stitt JA, Thomadsen BR, Buchler DA. The adverse effect of treatment prolongation in cervical carcinoma. Int J Radiat Oncol Biol Phys. 1995 Jul 30;32(5):1301-7. doi: 10.1016/0360-3016(94)00635-X. PMID 7635769
- [Background] Begg AC, Hofland I, Van Glabekke M, et al. Predictive value of potential doubling time for radiotherapy of head and neck tumor pa- tients: results from the EORTC cooperative trial 22851. Semin Radiat Oncol 1992;2:22-25.
- [Background] Kim YS, Choi EK, Lee JS et al. Consolidation chemotherapy with monthly Paclitaxel and Cisplatin (PC) or observation after concurrent chemoradiotherapy for locally advanced non-small cell lung cancer (NSCLS): randomized phase II study. J Thorac Oncol 2007; 2:449s.
- [Background] Huber R, M, Engel-Riedel W, Kollmeier J et al. GILT study: oral vinorel- bine (NVBo) and cisplatin (P) with concomitant radiotherapy (RT) fol- lowed by either consolidation (C) with NVBo plus P plus best supportive care (BSC) or BSC alone in stage (st) III non-small cell lung cancer (NSCLC): final results of a phase (ph) III study. J Clin Oncol 2012;30: 452s (suppl, abstr 7001).
- [Background] Ahn JS, Ahn YC, Kim JH, Lee CG, Cho EK, Lee KC, Chen M, Kim DW, Kim HK, Min YJ, Kang JH, Choi JH, Kim SW, Zhu G, Wu YL, Kim SR, Lee KH, Song HS, Choi YL, Sun JM, Jung SH, Ahn MJ, Park K. Multinational Randomized Phase III Trial With or Without Consolidation Chemotherapy Using Docetaxel and Cisplatin After Concurrent Chemoradiation in Inoperable Stage III Non-Small-Cell Lung Cancer: KCSG-LU05-04. J Clin Oncol. 2015 Aug 20;33(24):2660-6. doi: 10.1200/JCO.2014.60.0130. Epub 2015 Jul 6. PMID 26150444
- [Background] Tsujino K, Kurata T, Yamamoto S, Kawaguchi T, Kubo A, Isa S, Hasegawa Y, Ou SH, Takada M, Ando M. Is consolidation chemotherapy after concurrent chemo-radiotherapy beneficial for patients with locally advanced non-small-cell lung cancer? A pooled analysis of the literature. J Thorac Oncol. 2013 Sep;8(9):1181-9. doi: 10.1097/JTO.0b013e3182988348. PMID 23883782
- [Derived] Qiu B, Xi Y, Liu F, Li Y, Xie X, Guo J, Guo S, Wu Y, Wu L, Liang T, Ding Y, Zhang J, Wu Q, Liu H. Gut Microbiome Is Associated With the Response to Chemoradiotherapy in Patients With Non-small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2023 Feb 1;115(2):407-418. doi: 10.1016/j.ijrobp.2022.07.032. Epub 2022 Jul 26. PMID 35905860
- [Derived] Chen N, Li Q, Wang S, Xiong M, Luo Y, Wang B, Chen L, Lin M, Jiang X, Fang J, Guo S, Guo J, Hu N, Ai X, Wang D, Chu C, Liu F, Long H, Wang J, Qiu B, Liu H. Hypo-fractionated radiotherapy with concurrent chemotherapy for locoregional recurrence of non-small cell lung cancer after complete resection: A prospective, single-arm, phase II study (GASTO-1017). Lung Cancer. 2021 Jun;156:82-90. doi: 10.1016/j.lungcan.2021.04.020. Epub 2021 Apr 27. PMID 33933895